CLINICAL TRIAL: NCT04826991
Title: Wells and Enteric Disease Transmission - A Randomized Trial of Children Supplied Drinking Water From Private Wells (WET-Trial)
Brief Title: Wells and Enteric Disease Transmission
Acronym: WET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Heather Murphy, Adjunct Associate Research Professor, Temple University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25665-A (Full Trial); R01AI153376-01 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Diarrhea; Gastrointestinal Infection; Respiratory Viral Infection; Waterborne Diseases
Keywords: drinking water; private wells; UV disinfection
MeSH Terms: conditions — Diarrhea; Waterborne Diseases

STUDY DESIGN:
Intervention Model Description: A whole-home UV water treatment system will be installed and operated at a minimum of 50 millijoules per square centimeter.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, device installers, investigators, and outcomes assessor will all be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active UV Device (Active Comparator): A household water treatment device with a lamp emitting germicidal UV. The device will be operated at 50 millijoule per square centimeter to treat >99.9% of all bacteria, protozoa, and most viruses in water supplies.
  Interventions: Device: Active UV Device
- Inactive UV Device (Sham Comparator): A household water treatment device with a lamp not emitting germicidal UV but still emitting light (appears identical to the active UV device).
  Interventions: Device: Inactive UV Device

INTERVENTIONS:
Device: Active UV Device — Active water treatment system
  Arms: Active UV Device
Device: Inactive UV Device — Inactive water treatment system
  Arms: Inactive UV Device

SUMMARY:
Approximately 40 million people in the US are served by private, and frequently untreated, wells. Our best estimate is that 1.3 million cases of gastrointestinal illnesses (GI) per year are attributed to consuming water from untreated private wells in the US, but in reality, there are no robust epidemiological data that can be used to estimate cases of GI attributable to these sources. We propose the first randomized controlled trial (RCT) to estimate the burden of GI associated with private well water. We will test if household treatment of private well water by ultraviolet light (UV) vs. sham (inactive UV device) decreases the incidence of GI in children under 5. We will also examine the presence of viral, bacterial, and protozoan pathogens in stool and well water from participants. These data will fill a knowledge gap on sporadic GI associated with federally-unregulated private water supplies in the US.

DETAILED DESCRIPTION:
Investigators will conduct a triple-blinded randomized controlled trial of a whole-home UV water treatment device in southeastern Pennsylvania. Participating families will be randomized to receive an active UV device or a sham (inactive) UV device. Following the installation of the device, participants will be followed for one year. During that year, participants will respond to weekly text messages to report the presence of symptoms associated with gastrointestinal and respiratory illness in their children. Upon reporting symptoms, participants will complete an illness questionnaire on details regarding the illness and other potential exposure events. A subset of participants will submit groundwater samples as well as stool and saliva samples from their children. Water and stool samples will be analyzed for common waterborne pathogens. Saliva samples will be analyzed for immunoconversions to common waterborne pathogens (exploratory aim).

Under the guidance of an interdisciplinary advisory committee we will execute the following aims:

Aim 1- Quantify the incidence rate of endemic childhood GI associated with consuming untreated private well water and compare that to the incidence rate of consuming well water treated by UV.

Aim 1a- Construct a Quantitative Microbial Risk Assessment (QMRA) using water quality data we collect to estimate the risk of childhood GI associated with consuming untreated private well water and compare the incidence from the risk model to the incidence we calculate in Aim 1.

Aim 2- Identify, quantify and compare viral, bacterial and protozoan pathogens in stool of children consuming UV treated or untreated (sham) private well water (including both asymptomatic and symptomatic cases).

Aim 3- Explore the presence of pathogens in untreated well water and stool samples of children consuming untreated private well water (sham group only).

ELIGIBILITY:
Inclusion Criteria:

* Child resides in Adams, Berks, Bucks, Carbon, Chester, Columbia, Cumberland, Dauphin, Delaware, Lackawanna, Lancaster, Lebanon, Lehigh, Luzerne, Monroe, Montgomery, Montour, Northumberland, Northampton, Perry, Pike, Schuylkill, Wayne, Wyoming, and York county in Pennsylvania and all counties in New Jersey.
* Household is served by a private well
* Participant child is under the age of 5 (under 4 at time of enrollment), who is a full-time resident of the home and drinks untreated well water
* Parent/guardian has access to a phone with texting capabilities

Exclusion Criteria:

* Child participant is immunocompromised
* Child participant has a chronic gastrointestinal condition
* Child takes daily oral steroids
* Household treats water for microbiological contamination before consumption
* Child exclusively drinks bottled water

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 908 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incident gastrointestinal illness | 12 months
  The investigators will collect data on the presence of gastrointestinal illness symptoms through weekly text messages. Households that report symptoms through text messages will be directed to an online illness questionnaire to characterize the symptoms (type, incidence, severity, duration, etc.), as well as relevant exposure information such as recent travel, exposure to ill persons, etc. Incident gastrointestinal illness (GI) is defined by the reporting of a minimum of three episodes of diarrhea or vomiting in a 24 hour period. Each illness will be considered distinct when separated by ≥ 6 symptom-free days.

SECONDARY OUTCOMES:
Acute respiratory infection | 12 months
  The investigators will collect data on the presence of acute respiratory infection symptoms through weekly text messages. Households that report symptoms through text messages will be directed to an online illness questionnaire to characterize the symptoms (type, incidence, severity, duration, etc.) as well as relevant exposure information such as recent travel, exposure to ill persons, etc. Acute respiratory infection is defined by the reporting of nasal congestion/discharge, sore throat or mouth sores, or cough lasting at least one day, in the absence of another explanation, such as isolated cough without nasal symptoms in known reactive airways disease. Each illness will be considered distinct when separated by ≥ 6 symptom-free days.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Murphy, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee D, Denno D, Tarr P, Wu J, Stokdyk JP, Borchardt M, Murphy HM. Study design and methods of the Wells and Enteric disease Transmission (WET) Trial: a randomised controlled trial. BMJ Open. 2023 Mar 2;13(3):e068560. doi: 10.1136/bmjopen-2022-068560. PMID 36863739